CLINICAL TRIAL: NCT07077525
Title: Effect of Vildagliptin Versus Dapagliflozin as Add on Therapy to Metformin on Cardiovascular Risk Factors in Egyptian Type II Diabetic Obese Patients: Potential Impact of Genetic Polymorphism
Brief Title: Effect of Vildagliptin Versus Dapagliflozin as Add on Therapy to Metformin on Cardiovascular Risk Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Khalid Saber, Assistant Lecturer, Faculty of Pharmacy, Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE00302
Record Dates: First submitted 2025-06-24; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes mellitus; Vildagliptin; Dapagliflozin; Metformin; Cardiovascular risk factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin; Metformin; Vildagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin plus metformin (Active Comparator): 70 patients with T2DM: will be given metformin plus vildagliptin combination as per the standard of care in a physician's practice.
  Interventions: Combination Product: Dapagliflozin + Metformin
- Vildagliptin plus metformin (Active Comparator): 150 patients with T2DM: will be treated with metformin plus dapagliflozin combination as per the standard of care in a physician's practice.
  Interventions: Combination Product: Vildagliptin + Metformin

INTERVENTIONS:
Combination Product: Dapagliflozin + Metformin — 70 patients with T2DM were treated once daily with Dapa plus Met combination (Dapavildactin plus®, Liptis Pharmaceuticals, Egypt) in a dose titrated from 5 mg Dapa and 1000 mg Met up to a maximum of 10 mg Dapa and 2000 mg metformin as per the standard of care in a physician's practice
  Arms: Dapagliflozin plus metformin
Combination Product: Vildagliptin + Metformin — 126 patients with T2DM were treated with Vilda plus Met combination (Gliptus plus®, EVA pharma, Egypt ) in initial daily dose of 50 mg Vilda and 500 mg Met . The medication is titrated gradually up to Vilda 50 mg and metformin 1000 mg twice daily as per the standard of care in a physician's practice
  Arms: Vildagliptin plus metformin

SUMMARY:
The overarching hypothesis of this study is that vildagliptin (vilda) as add on therapy to metformin (met) in Egyptian type 2 diabetic obese patient will produce an equal, if not better, glycemic control and will reduce cardiovascular risk factors compared to dapagliflozin (dapa). However, there are interindividual differences in response to vildagliptin among Egyptian population which might be due to gender difference and/ or mutation in one or more of the DDP-4 gene, GLP1 receptor gene and KATP channel gene. These potential differences could favor pharmacogenomic selection of candidate patient.

Global aim of this study:

To compare effects of the DPP-4 inhibitor (vildagliptin) versus SGLT4 inhibiter (dapagliflozin) as add on therapy to metformin to control cardiovascular risk factors in Egyptian obese patients with type 2 diabetes and furthermore to investigate the possible interindividual variation to vildagliptins response.

Specific aims:

Evaluation of efficacy and safety of vildagliptin plus metformin versus dapagliflozin plus metformin in Egyptian obese patients with type 2 diabetes mellitus (T2DM).

Examining of interindividual difference in hypoglycemic response to the used treatment arms among participants of the study.

Assessment of response in relation to sex difference in Egyptian population. Investigation of vasculoprotective effects of different treatment with special emphasis on atherogenesis.

Investigating the efficacy of different treatment in controlling individual cardiovascular risk factors in preventing or slowing atherosclerotic cardiovascular diseases in people with diabetes Exploring of whether genetic variation in the DPP4 gene, GLP1 receptor and KATP channel affects incretin levels, insulin secretion, and glucose tolerance in participants of the study.

Examining the associations between genetic variations of DPP-4 gene in men and women involved in this study

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a metabolic disorder resulting from a defect in insulin secretion, insulin action, or both. It is characterized by chronic hyperglycemia and is associated with a heavy health burden and macrovascular complications.

Because of the associated microvascular and macrovascular disease, diabetes accounts for almost 14% of United States health care expenditures, at least one-half of which are related to complications such as myocardial infarction, stroke, end-stage renal disease, retinopathy, and foot ulcers .

Common conditions coexisting with T2DM (e.g., hypertension and dyslipidemia) are clear risk factors for atherosclerotic cardiovascular diseases (ASCVD). Numerous studies have shown the efficacy of controlling individual cardiovascular risk factors in preventing or slowing ASCVD in people with diabetes. Furthermore, there is evidence that measures of 10-year coronary heart disease (CHD) risk among U.S. adults with diabetes have improved significantly over the past decade and that ASCVD morbidity and mortality have decreased . Thus, cardiovascular risk factors should be systematically assessed at least annually in all patients with diabetes. These risk factors include duration of diabetes, obesity/overweight, hypertension, dyslipidemia, smoking, a family history of premature coronary disease, chronic kidney disease, and the presence of albuminuria. Modifiable abnormal risk factors should be treated as described in the guidelines .

The general goals of the treatment of DM are to provide glycemic control, avoid acute complications, prevent, or delay the appearance of chronic complications of the disease, and thus to improve the quality of life. The management of type 2 DM also includes managing conditions associated with T2DM, such as obesity, hypertension, dyslipidemia, and cardiovascular disease. Initial treatment of T2DM includes both pharmacologic and non-pharmacologic therapy (lifestyle modification) for all patients. First-line therapy depends on comorbidities, patient-centered treatment factors, and management needs and generally includes metformin and comprehensive lifestyle modification. Other medications such as sulfonylureas, Dipeptidyl-peptidase 4 (DPP-4) inhibitors, glucagon-like peptide 1 receptor agonists (GLP1), sodiumglucose cotransporter 2 inhibitors (SGLT2), are usually added to metformin based on glycemic needs for individuals with T2DM with or at high risk for ASCVDs, heart failure, and/or chronic kidney disease.

Metformin is effective, safe, inexpensive, and may reduce risk of cardiovascular events and death. In addition, metformin is available in an immediate-release form for twice-daily dosing or as an extended-release form that can be given once daily. The latest challenge to the place of metformin has come from the recent demonstration of substantial cardiovascular outcomes benefits with GLP-1 receptor agonists and SGLT2 inhibitors.

Based in clear evince from large-scale randomized trials documenting important benefits of SGLT2 inhibitors to cardiovascular system and kidney, these agents are now recommended as the preferred second-line therapy in people who do not achieve sufficient glucose control on metformin alone, particularly for those with heart failure or chronic kidney disease . Furthermore, new guidelines from the European Society of Cardiology, developed in collaboration with the European Association for the Study of Diabetes, suggest that SGLT2 inhibitors be used in patients with T2DM who are at high or very high cardiovascular risk, irrespective of whether they are treatment-naïve or already receiving metformin .

Vildagliptin is a representative of Dipeptidyl Peptidase-4 (DPP-4) inhibitors, antihyperglycemic drugs, approved for use as monotherapy and combination therapy in type 2 diabetes mellitus. By inhibiting enzymatic decomposition, DPP-4 inhibitors increase the half-life of incretins such as GLP-1 and GIP and prolong their action. Interestingly, some studies present promising results suggesting the anti-sclerotic and vasculoprotective effects of vildagliptin. Vildagliptin can limit inflammation by suppression of the NF-κB (nuclear factor kappa-light-chain-enhancer of activated B cells) signaling pathway and proinflammatory agents such as TNF-α (tumor necrosis factor α)and IL-8 (Interleukin 8). This DPP-4 inhibitor also reduces macrophage foam cell formation, which plays a key role in atheromatous plaque formation and stability. The reasons for the good response and cardio-protective effects of DDP-4 inhibitor drugs are largely unknown. In addition, there is no detailed study on Egyptian obese patients with type 2 diabetes comparing vildagliptin to dapagliflozin concerning controlling cardiovascular risk factors and still all available guidelines prefer use of SGLT2 inhibitors over DDP-4 inhibitors for type 2 diabetic patients with ASCVD or risk, these might be due to lacking sufficient evidence about cardiovascular protective benefits of DDP-4 inhibitors.

Importantly, one relevant DPP-4 substrate, besides glucagon-like peptide-1 (GLP-1), is stromal cell derived factor 1α (SDF-1α). SDF-1∝ may act as a double edge sword with respect to the CV system . It is a potent chemokine stimulating stem cell mobilization from the bone marrow and, it plays a positive role in the angiogenic process following acute ischemic injury. On the other hand, SDF-1α has recently emerged as a robust biomarker of CV diseases and mortality whereas higher SDF-1α levels were associated with the presence of several CV risk factors and independently with heart failure and with 10-year all-cause mortality. Furthermore, in the chronic renal insufficiency cohort study, higher SDF-1∝ levels predicted increased 6-year mortality. Based on these contradictory data it was pertinent to explore the real effect of DDP-4 inhibitor in comparison to already stablished benefits of SGLT2 inhibitors.

Of particular interest, Inter-individual variance in the responsiveness to DPP-4 inhibitors was reported. A common variant, i.e., SNP rs6741949, in the DPP4 gene interacts with body adiposity and negatively affects glucose-stimulated GLP-1 levels, insulin secretion, and glucose tolerance. Another variants rs6923761 in GLP1 receptor gene and rs2285676 in KATP channel gene might also affect the effect to Vildagliptin. Whether this SNP underlies the potential inter-individual variance in responsiveness to DPP-4 inhibitors, at least in subjects with high body fat content, remains to be another hot topic to be addressed to tailor the therapeutic option with vildagliptin to the right patient.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria involve Egyptian patients with newly documented T2DM diagnosis (naïve)
* 40-60 years old
* HbA1c level between 6.5% - 10.0% (47.5-107.7 mmol/mol) before study initiation
* obese (BMI ≥30 kg/m2)
* no history of established CV disease
* ability to understand and to sign a written informed consent document
* outpatients
* TSH and liver function within normal limit and no evidence of kidney diseases.

Exclusion Criteria:

* Diagnosis of T1DM
* subjects with any serious medical condition requiring hospitalization
* subjects with unstable cardiac disorders such as heart failure, refractory angina, uncontrolled arrhythmias, critical valvular heart disease and severe uncontrolled hypertension
* renal or liver failure
* females of childbearing potential or who are pregnant
* breast-feeding
* subjects using any drug that could interfere with the glucose level (e.g. systemic corticosteroids) and participation in any other clinical trial.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of HbA1c level | 0,6 and 12 months of treatment
  Measurement of serum levels of HbA1C as a percentage (%) at 0 (baseline) 6 and 12 months. Change of serum level of HbA1C due to treatments after 12 months and determine the frequency of participants achieved reduction of HbA1c level by more than 1%
Evaluation of serum level of FBG | 0, 6 and 12 months
  Measurement of serum level of FBG as (mg/dl) at 0,6 and 12 months. Change of serum level of FBG due to treatments after 12 months
Evaluation of serum level of PPG | 0.6 and 12 months
  Measurement of serum level of PPG as (mg/dl) at 0,6 and 12 months. Change of serum level of PPG due to treatments after 12 months

SECONDARY OUTCOMES:
Evaluation of Body mass index (BMI) | 0,6 and 12 months of treatment
  Change in body mass index (kg/m2) due to different treatments from baseline to 6, and 12 months.
Evaluation of serum inflammatory cytokines | 0 and 12 months of treatment
  Assessment of serum level of interleukin 8 (IL8), nitric oxide (NO) and tumor necrosis factor subtype alpha (TNF-α) at baseline and 12-months post treatment
Assessment of genetic variation | After 12 months of treatment
  Genotyping assays among participant of study and its relation to glycemic control and other cardiovascular risk factors for certain genes SNP rs6741949 in the DPP4 gene, SNP rs6923761 in the GLP1 receptor and SNP rs2285676, in the KATP gene.
Assessment of lipid profile parameters | 0, 6 and 12 months of treatment
  Measurement of lipid profile parameters at 0 (baseline) 6 and 12 months. Change of lipid profile parameters due to different treatments from baseline to 12 months of treatment
Assessment of a common variant, SNP rs6741949, in the DPP4 gene | After 12 months of treatment
  Assessment of a common variant, SNP rs6741949, in the DPP4 gene to determine the highest frequency and responsive alleles
Assessment of a common variant SNP rs6923761, in the GLP1 receptor | After 12 months of treatment
  Assessment of a common variant SNP rs6923761, in the GLP1 receptor to determine the highest frequency and responsive allele.
Assessment of a common variant, SNP rs2285676, in the KATP gene. | After 12 months of treatment
  Assessment of a common variant, SNP rs2285676, in the KATP gene to determine the highest frequency and responsive allele.

OTHER OUTCOMES:
Measurement of homocysteine and vitamin B12 serum levels | 0 and 12 months
  . Assessment of homocysteine and vitamin b12 was in serum at 0 and 12 months
Measurement of stromal cell derived factor and vascular cell adhesion molecule 1 in serum | 0 and 12 months of treatment
  Serum level of stromal cell derived factor 1 alpha (SDF-1α) as a biomarker of CV risk and mortality was determined at 0 and 12 months
Evaluation of serum liver biomarkers | 0, 6 and 12 months of treatment
  Serum liver biomarkers [alanine aminotransferase (ALT), aspartate aminotransferase (AST), direct and total bilirubin] will be assessed using standard colorimetric techniques
Assessment of serum creatinine (sCr) | 0 and 12 months of treatment
  Measurement of serum creatinine (mg/dl) at 0 and 12 months of treatment to determine the change of serum creatinine due to different treatments from baseline to 12 months of treatment
Measurement of albumin/creatinine ratio | 0 and 12 months of treatment
  Measurement of albumin/creatinine ratio (mg/g) at 0 and 12 months of treatment to determine the change of A/c ratio due to different treatments from baseline to 12 months of treatment
Assessment of eGFR | 0 and 12 months of treatment
  Measurement of eGFR (ml/min) at 0 and 12 months of treatment to determine the change of eGFR due to different treatments from baseline to 12 months of treatment
Assessment of CrCl | 0 and 12 months of treatment
  Measurement of CrCl (ml/min) at 0 and 12 months of treatment to determine the change of CrCl due to different treatments from baseline to 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Khalid S Hassanien, Assistant lecturer, Principal Investigator — al-azhar university, faculty of pharmacy, cairo.; Memy M Hegazy, professor, Study Director — al-azhar university, faculty of pharmacy, cairo.; Atef A Bassyouni, Profepssor, Study Chair — Medical consultant . National Institute of Diabetes and Endocrinology; Raed S Ismail, Professor, Study Chair — al-azhar university, faculty of pharmacy, cairo.; Mohammed F Elshafie, Assistant professor, Study Chair — al-azhar university, faculty of pharmacy, cairo.
Locations (1):
- Al-Azhar university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
We will report the results without disclosing patients personal information or images for human ethical protection reasons and culture habits